CLINICAL TRIAL: NCT00061399
Title: Prospective Memory in Normal and Head-Injured Children
Brief Title: Prospective Memory in Children With Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: K23HD040896 (NIH)
Record Dates: First submitted 2003-05-27; First posted 2003-05-28 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2007-04

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Prospective memory
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Prospective memory (PM) is memory to complete future tasks, such as recalling to give a note to someone when you next see them, pick up milk on the way home, or remembering to keep an appointment. This study will evaluate PM in children with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
While much has been learned about how children with TBIs learn and recall stories, word lists, and pictures, little is known about how they perform PM tasks. Impairment in PM could have serious implications for academic and vocational pursuits. This study will investigate PM in children with mild or severe TBI. The study will focus on three major themes: 1) strategies that may help children with TBI overcome or minimize their PM deficits; 2) how specific areas of cognition can be impaired following TBI and in turn impair PM; and 3) the impact of PM deficits on a child's daily functioning, both at school and at home. The study will also evaluate children without TBI (control group).

Each child will participate in one study evaluation. The evaluation will last approximately 4 hours, with a lunch break and other rest breaks as necessary. Assessments will include neuropsychological tests of attention, memory, and general intellectual functioning. Experimental tasks will include measures of metacognition for prospective memory, elucidation of strategic versus automatic processes involved in PM, and the effect of motivation manipulations in overcoming PM deficits with varying working memory loads. The child's parent or guardian will also be asked to complete some tests to measure the impact of PM deficits on the child's daily home life.

ELIGIBILITY:
Inclusion Criteria

* English speaker
* Minimum birth weight of 2500 grams (5.5 lbs) and 37 weeks' gestation

Additional Inclusion Criteria for Children with Traumatic Brain Injury

* Head injury resulting in a post-resuscitation Glasgow Coma Scale score of either 13 to 15 or 3 to 8
* No evidence of hypoxic injury

Exclusion Criteria

* History of epilepsy, mental retardation, or documented evidence of developmental dysfunction
* Previous hospitalization for head injury involving loss of consciousness or post-concussional symptoms
* History of autism, major psychiatric disorder, or pervasive developmental delay
* History of meningitis or encephalitis
* History of child abuse
* History of chronic or uncontrolled serious physical disorders (cancer, uncontrolled diabetes, cystic fibrosis, etc.)
* Note: siblings of participants with TBI or orthopedically-injured comparison children will not be enrolled to maintain the independence of the groups

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 178
Dates: Start 2002-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. McCauley, Ph.D., Principal Investigator — Baylor College of Medicine